CLINICAL TRIAL: NCT04660396
Title: Monitoring Outpatient Blood VolumE in Heart Failure
Acronym: MOVE-HF
Status: Completed | Type: Observational
Sponsor: Daxor Corporation (Industry)
Collaborators: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MOVE-HF
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
Keywords: Plasma Volume; Red Blood Cell Volume; Blood Volume; Diuresis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Outpatients following discharge for treatment of heart failure: Daxor Corporation's commercially available Blood Volume Analyzer, BVA-100, will be performed at 5 timepoints for each patient.
  Interventions: Device: BVA-100

INTERVENTIONS:
Device: BVA-100 — The BVA-100 is a software package designed to calculate human blood volume using the method of tracer dilution. It uses tagged serum albumin (a commonly used tag is 131I, resulting in "131I -HSA"). Data inputs to the software come from the measured characteristics of subject blood samples (hematocrit and tracer concentration) and tracer calibration standards. The package also calculates the subject expected (or ideal) blood volume from physical parameters. Hyper- or hypovolemia, associated red blood cell volumes, and transudation rate are reported, with statistics showing the quality of the results. The subject blood samples and calibration standards are measured in a gamma counter, whose output is automatically, or manually, input to this calculation program.

SUMMARY:
In patients discharged following heart failure treatment, the consistency of blood volume status and components over time is unknown. The primary objective is to describe the rate of change, if any, of the plasma volume and red blood cell volume following hospitalization and discharge of patients with heart failure.

DETAILED DESCRIPTION:
Over 6 million Americans suffer from heart failure, one of the most prevalent and deadly diseases. High 30-day readmission and mortality rates have persisted despite advances in care. Clinical guidelines suggest blood volume assessment and clinical management to euvolemia or normal blood volume, but standard methods of blood volume diagnosis have been shown to be unreliable. FDA-cleared Blood volume analysis (BVA) has been used to quantify otherwise undiagnosed blood volume derangements in heart failure and other indications. Also, care guided by BVA has been demonstrated to improve inpatient heart failure readmission and mortality. A similar analysis has not previously been performed immediately following hospital discharge, though this period is understood to be challenging due to high variability of patient status, physiology, and compliance.

This is a prospective, single-center, observational open-label study. The primary objective is to quantify changes to plasma volume and red blood cell volume over a 12 week period post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male and female patients with primary or secondary admission diagnosis of acute heart failure exacerbation
* > 18 years of age
* Able and willing to provide consent
* Reduced or preserved LVEF

Exclusion Criteria:

* Diagnosed with current acute strokes
* Pregnant women
* Severe hypotension requiring resuscitation, intubation or circulatory support
* Cardiogenic shock
* Patients with known cardiac amyloid and hypotension
* Known allergy to iodine or iodinated albumin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to Geisinger Medical Center with a diagnosis of acute heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Quantify volume shifts in post discharge heart failure patients | 12 weeks
  Accurately quantify changes to plasma volume and red blood cell volume in HF outpatients over the 12-week period following discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carry, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No